CLINICAL TRIAL: NCT07246564
Title: An Open-label, Prospective, Single-arm Study Assessing the Efficacy and Safety of Rozanolixizumab in Adult Chinese Participants With Generalized Myasthenia Gravis
Brief Title: Phase 4 Study Evaluating Efficacy and Safety of Rozanolixizumab in Adult Chinese Participants With Generalized Myasthenia Gravis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG0033
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Myasthenia Gravis
Keywords: Rozanolixizumabg, gMG
MeSH Terms: conditions — Myasthenia Gravis | interventions — rozanolixizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rozanolixizumab (Experimental): Participants will receive 6 dose per cycle of subcutaneous infusion of rozanolixizumab
  Interventions: Drug: Rozanolixizumab

INTERVENTIONS:
Drug: Rozanolixizumab — Subcutaneous infusion

SUMMARY:
The purpose of the study is to assess the clinical efficacy of rozanolixizumab in adult Chinese participants with generalized myasthenia gravis (gMG) in the first Treatment Cycle.

ELIGIBILITY:
Inclusion Criteria:

* Study participant must be ≥18 years of age at the time of signing the informed consent form (ICF)
* Study participant has documented diagnosis of generalized myasthenia gravis (gMG) at the Screening Visit based on study participant's history and supported by previous evaluation
* Study participant has a confirmed positive record of autoantibodies against acetylcholine receptor (AChR) or muscle-specific kinase (MuSK) documented in the medical history at the Screening Visit
* Study participant has Myasthenia Gravis Foundation of America (MGFA) Clinical Classification II to IV at Screening Visit.
* Study participant with a myasthenia gravis-activities of daily living (MG-ADL) score of at least 3 points from non-ocular symptoms and a quantitative myasthenia gravis (QMG) score of at least 11 at the Screening and Baseline visits in the first Treatment Cycle.
* Study participant is considered for additional treatment by the investigator
* Body weight ≥35kg at the Screening Visit

Exclusion Criteria:

* Study participant has a known hypersensitivity to any components of the study drug or any other anti-neonatal Fc receptor (anti-FcRn) medications
* Study participant has a clinically important active infection including unresolved or not adequately treated infection in the opinion of the investigator
* Study participant with a known tuberculosis (TB) infection, at high risk of acquiring TB infection, or latent tuberculosis infection (LTBI), or current/history of nontuberculous mycobacterial infection (NTMBI)
* Study participant has previously received rozanolixizumab drug product
* Study participant has received any vaccine in the 4 weeks prior to the initiation of rozanolixizumab treatment or intends to receive any vaccine within 2 weeks after the last infusion of rozanolixizumab. Note: For participants that are on rozanolixizumab treatment, vaccination with live or live-attenuated vaccines is not recommended. During the whole study period, all other vaccines should take place at least 2 weeks after the last infusion of a Treatment Cycle and 4 weeks before initiating the next cycle
* Study participant has been treated with prohibited immunosuppressants, biologics, and other therapies within the timeframe shorter than the treatment-free period
* Study participant with severe (defined as Grade 3 on the MG-ADL scale) weakness affecting oropharyngeal or respiratory muscles, or who has myasthenic crisis or impending crisis. Note: Impending Crisis is defined as bulbar or respiratory symptoms of a patient who significantly worsens in a short time (≤2 weeks) and meet MGFA IVb or score 3 in one QMG bulbar muscle item, or score 2 in respiratory muscle item, or bulbar+respiratory items score ≥4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-10-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Day 43 in Myasthenia Gravis-Activities of Daily Living (MG-ADL) score in the first Treatment Cycle | Baseline to Day 43 (in first treatment cycle)
  The total MG-ADL score is obtained by summing the responses to each individual item (8 items; Grades: 0, 1, 2, 3). The score ranges from 0 to 24, with a higher score indicating more disability.
  A positive change indicates worsening and a negative change indicates improvement.

SECONDARY OUTCOMES:
MG-ADL responder (≥2.0-point improvement from Baseline) at Day 43 in the first Treatment Cycle | Baseline to Day 43 (in first treatment cycle)
  A MG-ADL responder is defined as achieving at least 2.0-point improvement in the MG-ADL total score from Baseline.
Change from Baseline to Day 43 in Myasthenia Gravis-Composite (MG-C) score within first 6 week treatment cycle | Baseline to Day 43 (in first treatment cycle)
  The MG-C scale is a validated assessment, with a higher score indicating more severe disease and a 3-point change being of clinical relevance. The scale tests 10 items, with individual items being weighted differently. The overall score ranges from 0 to 50 (more severe disease).
  The items included ptosis/upward gaze (range: 0 [>45 second] - 3 [Immediate]), double vision on lateral gaze (range: 0 [>45 second] - 4 [Immediate]), eye closure (range: 0 [Normal] - 2 [severe weakness]), talking (range: 0 [Normal] - 6 [difficult to understand speech]), chewing (range: 0 [Normal] - 6 [gastric tube]), swallowing (range: 0 [Normal] - 6 [gastric tube]), breathing (range: 0 [Normal] - 9 [ventilator dependence]), neck flexion (range: 0 [Normal] - 4 [severe weakness]), shoulder abduction (range: 0 [Normal] - 5 [severe weakness]) and hip flexion (range: 0 [Normal] - 5 [severe weakness]), lower scores= lower disease activity.
Change from Baseline to Day 43 in Quantitative Myasthenia Gravis (QMG) score within first 6-week treatment cycle | Baseline to Day 43 (in first treatment cycle)
  The total QMG score is obtained by summing the responses to each individual item (13 items [ocular and facial involvement, swallowing, speech, limb strength, and forced vital capacity]; Responses: None=0, Mild=1, Moderate=2, Severe=3). The QMG is a validated assessment, with a higher score indicating more severe disease. Scoring for each item ranges from no weakness (0) to severe weakness (3), with an overall score range from 0 to 39. A 3-point change in the total score is considered clinically relevant.
Change from Baseline to Day 43 in Myasthenia Gravis (MG) Symptoms Patient Reported Outcome (PRO) 'Muscle Weakness Fatigability' score within first 6-week treatment cycle | Baseline to Day 43 (in first treatment cycle)
  The MG symptoms PRO instrument consisted of 42 items across 5 scales: ocular muscle weakness (items 1-5); bulbar muscle weakness (items 6-15); respiratory muscle weakness (items 16-18); physical fatigue (items 19-33) and muscle weakness fatigability (items 34-42). Study participants will be asked to choose response option that best describes how frequently they experienced muscle weakness fatigability (items 34-42) over the past 7 days using a 5-point Likert scale (1="none of the time" to 5="all of the time") for each item.
Change from Baseline to Day 43 in MG Symptoms PRO 'Physical Fatigue' score within first 6-week treatment cycle | Baseline to Day 43 (in first treatment cycle)
  The MG symptoms PRO instrument consisted of 42 items across 5 scales: ocular muscle weakness (items 1-5); bulbar muscle weakness (items 6-15); respiratory muscle weakness (items 16-18); physical fatigue (items 19-33) and muscle weakness fatigability (items 34-42). Study participants will be asked to choose the response option that best describes how frequently they experienced physical fatigue (items 19-33) over the past 7 days using a 5-point Likert scale (1="none of the time" to 5="all of the time") for each item.
Percentage of participants with treatment-emergent adverse events (TEAEs) | Up to End of study (40 weeks)
  Treatment Emergent Adverse Events (TEAEs) are any untoward medical incidence in a participant after the administration of study treatment, whether or not these events are related to study treatment.
Percentage of participants with TEAEs leading to withdrawal of investigational medicinal product (IMP) | Up to End of study (40 weeks)
  Treatment Emergent Adverse Events (TEAEs) are any untoward medical incidence in a participant after the administration of study treatment, whether or not these events are related to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 22733 (UCB)
Locations (6):
- China (6):
  - Mg0033 20295, Changsha
  - Mg0033 20348, Fuzhou
  - Mg0033 20185, Jinan
  - Mg0033 20172, Shanghai
  - Mg0033 20184, Shenzhen
  - Mg0033 20204, Suzhou

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org